CLINICAL TRIAL: NCT00067223
Title: Bi-hemispheric Plasticity Elicited By Unilateral Finger Motor Training
Brief Title: Studying Use-Dependent Plasticity
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030273; 03-N-0273
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-06-25

CONDITIONS: Healthy
Keywords: Transcranial Magnetic Stimulation (TMS); Unilateral Finger Movement; Interhemispheric Inhibition; Motor Training; Plasticity; Healthy Volunteer; HV

SUMMARY:
Recent studies suggest that when patients learn a new motor movement, it may cause a change in the way the nerves act in the area of the brain that controls that movement. This change is called use-dependent plasticity.

The purpose of this study is to determine the direction and extent of the changes that take place in the brain areas that control movement in the untrained finger after the training of the opposite finger. The study outcomes may help researchers to develop rehabilitation strategies for people who have suffered brain injuries.

Eighteen healthy adults age 18 years or older will be enrolled in this study. Participants will undergo a clinical exam and then come back to the Clinical Center three times for sessions that will last approximately 2 hours each. For each session, participants' forearms will be immobilized and a small electronic device will be attached to each index finger so that researchers can measure their movements. Participants will be asked to move either index finger and to observe and concentrate on its movement. Investigators will perform transcranial magnetic stimulation (TMS) before and after these motor exercises. For TMS, a wire coil is held over the scalp and a brief electrical current passes through the coil, creating a magnetic pulse that electrically stimulates the brain.

DETAILED DESCRIPTION:
Motor training consisting of repetition of unilateral finger movements leads to use-dependent plasticity (UDP) in the contralateral primary motor cortex, M1, in normal volunteers. It is conceivable that motor training in one hand, in addition to changes in the contralateral M1, could elicit plastic changes in the ipsilateral M1. The purpose of this study is to test this hypothesis: Training consisting of repetition of a unilateral finger movement elicits plastic changes in the cortical representation of the homonymous untrained finger in the ipsilateral M1. The study will be performed on normal volunteers and will consist of three to five separate training sessions. The endpoint measure will be, for each session, the change in the direction of the movements evoked by TMS in the untrained index finger as a function of the opposite index finger.

ELIGIBILITY:
* INCLUSION CRITERIA:

Only healthy volunteers 18 years or older will be included in this protocol. Handedness will be assessed by the Edinburgh Inventory Scale. All experimental sessions will be studied on outpatient basis. Normal Volunteers with right-handedness will be eligible to participate.

EXCLUSION CRITERIA:

Subjects with the history of epilepsy, surgery with metallic implants or known history of metallic particles in the eye, cardiac pacemaker, neural stimulators, cochlear implants, history of drug abuse, psychiatric illness (depression), hypertension or use of medications that influence synaptic plasticity, will be excluded as evaluated by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-08-05; Study Completion 2007-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liepert J, Dettmers C, Terborg C, Weiller C. Inhibition of ipsilateral motor cortex during phasic generation of low force. Clin Neurophysiol. 2001 Jan;112(1):114-21. doi: 10.1016/s1388-2457(00)00503-4. PMID 11137668